CLINICAL TRIAL: NCT02562339
Title: Examining the Psychosocial Effects of Resiliency Training for Adolescents With Craniofacial Conditions and Their Caregivers
Brief Title: Resiliency Training for Adolescents With Craniofacial Conditions and Their Caregivers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the departure of study staff and lack of interest by potential subjects and the sponsor, the investigators decided to end the study.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Foundation For Faces of Children (Other)
Responsible Party: Principal Investigator, John W. Denninger, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015P000956
Record Dates: First submitted 2015-09-21; First posted 2015-09-29 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Craniofacial Abnormalities
MeSH Terms: conditions — Craniofacial Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMART-3RP for Parents or Caregivers (Experimental): Participants will receive an 8-week behavioral intervention which teaches stress management and psychological resiliency-enhancing skills.
  Interventions: Behavioral: SMART-3RP
- SMART-3RP for Adolescent Patients (Experimental): Participants will receive an 8-week behavioral intervention which teaches stress management and psychological resiliency-enhancing skills.
  Interventions: Behavioral: SMART-3RP

INTERVENTIONS:
Behavioral: SMART-3RP — 8-week group intervention teaching relaxation and psychological resiliency enhancing skills. Topics include the relaxation response, meditation, and yoga.

SUMMARY:
This is a prospective study that will examine psychosocial improvements among CF adolescents and caregivers going through the Stress Management and Resiliency Training - Relaxation Response Resiliency Program (SMART-3RP).

ELIGIBILITY:
Inclusion Criteria for Adolescent Patients:

1. Adolescents aged 14 to 22
2. English fluency and literacy
3. Diagnosis of a craniofacial condition by self report

Inclusion Criteria for Parents or Other Caregivers:

1. Must be 18 years of age and older
2. English fluency and literacy
3. Parent or caregiver of a child or young adult with a craniofacial condition

Exclusion Criteria:

1. Unable to benefit from the program due to cognitive, psychiatric or other reasons based on the opinion of the group leader
2. Unable or unwilling to sign the informed consent documents

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Quality of Life (WHOQOL-BREF) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The WHOQOL-BREF comprises of 26 items which measure the following broad domains: physical health, psychological health, social relationships, and environment. The WHOQOL-BREF is a shorter version of the original instrument that may be more convenient for use in large research studies or clinical trials.
The 14-Item Resiliency Scale (RS-14) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The RS-14 measures stress coping ability in the face of adversity.

SECONDARY OUTCOMES:
Satisfaction with Life (SWL) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The Satisfaction with Life (SWL) scale is a reliable and valid 5-item self-report measure of global life satisfaction. Responses are made on a 7-point scale with higher scores reflecting higher life satisfaction.
Perceived Stress Scale (PSS-10) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The PSS is a widely used psychological instrument for the measurement of the perception of stress. This 10-itam scale is designed to measure the degree to which situations in one's life are appraised, or considered stressful. The scores range from 0-40, with a higher score indicating higher perceived stress. Items were designed to detect how unpredictable, uncontrollable and overloaded respondents find their lives.
Measure of Current Status (MOCS-A) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The MOCS-A is a 13-item measure assessing participants' current self-perceived status on several skills such as: the ability to relax at will, recognize stress-inducing situations, restructure maladaptive thoughts, be assertive about needs, and choose appropriate coping responses as needed. Responses are made on a 7-point scale with higher scores reflecting higher life satisfaction.
Patient Health Questionnaire (PHQ) - caregivers only | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The PHQ measures symptoms of depression and functional impairment.
Patient Health Questionnaire for Adolescents (PHQ-A) - patients only | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  Symptoms of depression and functional impairment
Generalized Anxiety Disorder 7-item (GAD-7) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  A brief measure for assessing generalized anxiety disorder
Cognitive and Affective Mindfulness Scale (CAMS) - caregivers only | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The CAMS measures the degree to which individuals experience their thoughts and feelings.
Child and Adolescent Mindfulness Measure (CAMM) - patients only | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  Assesses mindfulness in children and adolescents
Interpersonal Reactivity Index (IRI) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The IRI assesses the cognitive and affective dimensions of empathy.
Distress Analogue Scales | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The Distress Analogue Scales measure participants' levels of stress, coping, distress, and discomfort.
The Gratitude Questionnaire (GQ-6) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The GQ-6 revised is a 6-item measure that assesses individual differences in the proneness to experience gratitude in daily life. Scores range from 6-42, with a higher score indicating a greater sense of gratitude.
Life Orientation Test (LOT) Optimism Scale | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The LOT Optimism Scale measures individual differences in generalized optimism versus pessimism.
Medical Outcomes Study (MOS) Social Support Survey | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The MOS Social Support Survey measures various dimensions of social support.
Rosenberg Self Esteem Scale (RES) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  Assesses levels of self esteem
The Body Image Quality of Life Inventory (BIQLI) - patients only | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  Measures patients' perception of their own body image and how it relates to quality of life.

OTHER OUTCOMES:
Age, Gender, Race, Ethnicity, Type of Craniofacial Condition, and Education Status of patients with craniofacial conditions and their caregivers | Baseline (week 0)
  This questionnaire asks patients/caregivers to report their age, gender, race, ethnicity, type of craniofacial condition, and highest level of education.
Expectancy Questionnaire | Baseline (week 0)
  Measures how much the participant believes the intervention will work
Intent to Attend Questionnaire | Baseline (week 0)
  On a scale from 1 ["Not likely" or "Not motivated"] to 3 ["Very likely" or "Very motivated"], participants are asked how likely and how motivated they are to attend the next session.
Participant Feedback - Program Satisfaction Questionnaire | Post-intervention (week 8)
  Measures how satisfied the participant is with the intervention

CONTACTS AND LOCATIONS:
Overall Officials: John W. Denninger, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States